CLINICAL TRIAL: NCT00934375
Title: A 28-Week Open Label Extension Study Evaluating Safety and Tolerability of Donepezil Hydrochloride in Subjects With Mild Cognitive Impairment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: James Prodafikas, Study Director, Eisai Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2020-A001-414
Record Dates: First submitted 2009-05-14; First posted 2009-07-08 (Estimated); Results first posted 2009-07-08 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2013-12

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Donepezil

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Aricept (donepezil hydrochloride)
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Aricept (donepezil hydrochloride) — 5 mg or 10 mg of donepezil hydrochloride (Aricept) taken orally once a day.
  Other Names: donepezil hydrochloride
  Arms: 1
Drug: placebo
  Arms: 2

SUMMARY:
This is a multi-center, open-label study of 28 weeks duration in subjects with Mild Cognitive Impairment who have completed the double-blind study (E2020-A001-412).

ELIGIBILITY:
Inclusion Criteria:

1. Age Range: Adult subjects (45 to 90 years of age inclusive)
2. Sex distribution: Men and women. Women of child-bearing potential (<1 year post menopausal) must be practicing effective contraception and have negative serum B-HCG at Screening. [Women who are breast-feeding are excluded.]
3. Subjects must have completed the one year, double-blind core trial (E2020-A001-412).
4. A completed Diagnostic Worksheet at the end of the double-blind core trial (E2020-A001-412) indicating no conversion to Alzheimer's Disease or dementia.
5. Health: Generally healthy and ambulatory or ambulatory-aided (i.e., walker or cane).
6. The subject must be expected to complete the entire study.
7. Subjects must be sufficiently fluent in English.
8. Subjects must have an informant who has daily contact with the subject (e.g., an average of 10 or more hours per week), can observe for possible adverse events and will accompany the subject to all visits.
9. Clinical laboratory values must be within normal limits, or if abnormal, judged clinically insignificant by the investigator (not likely to cause cognitive impairment or medical instability).

Exclusion Criteria:

1. Subjects who have not completed or have terminated early from the one year, double-blind core trial (E2020-A001-412).
2. Any subject without a completed diagnostic worksheet from Week 51 of the core double-blind trial (E2020-A001-412).
3. Any subject with a completed diagnostic worksheet from Week 51 of the core double-blind trial (E2020-A001-412) indicating conversion to Alzheimer's or other dementia.
4. Subjects with uncontrolled hypertension (sitting systolic >= 160mmHg and/or diastolic >=95mmHg) as assessed by the investigator, regardless of whether or not the subject is taking anti-hypertensive medications.
5. Subjects with a history of malignant neoplasms treated within five years prior to study entry (other than basal or squamous cell carcinoma of the skin); current evidence of malignant neoplasm; or recurrent or matastatic disease.
6. Subjects who have suffered a severe infection or a major surgical procedure within three months prior to baseline.
7. Subjects who may not be able to comply with the protocol.
8. Subjects with known hypersensitivity to piperidine derivatives or acetylcholinesterase(AChE)inhibitors.
9. Subjects with diabetes mellitis not controlled by diet and/or medication with a random serum glucose value of >170mg/dl.
10. Any condition which would make the subject, in the opinion of the investigator, unsuitable for the study.
11. Subjects who do not have a reliable informant (e.g., the informant has contact with the subject less than 10 hours per week).

Ages: 45 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2006-02; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anita Murthy, Study Director — Eisai Inc.
Locations (49):
- United States (49):
  - Neurology Neurodiagnostic Lab, LLC, Alabaster, Alabama
  - Pivotal Research Centers, Peoria, Arizona
  - Sun Health Research Institute, Sun City, Arizona
  - Northwest Neurospecialists, PLLC, Tucson, Arizona
  - The Neurology Center, Encinitas, California
  - Margolin Brain Institute, Fresno, California
  - Colaborative Neuroscience Network (CNS Network), Garden Grove, California
  - Nerve Pro Research, Irvine, California
  - Optimum Health Services, La Mesa, California
  - Pacific Research Network, San Diego, California
  - Neurological Research Institute, Santa Monica, California
  - CA Neuroscience Research, Sherman Oaks, California
  - Pacific Research Network, Vista, California
  - Yale University Alzheimers Disease Research Unit School of Medicine Department of Psychiatry, New Haven, Connecticut
  - North Broward Medical Center Memory Disorder Center, Deerfield Beach, Florida
  - Neurologic Consultants, Fort Lauderdale, Florida
  - Berma Research Group, Hialeah, Florida
  - Sunrise Clinical Research, Hollywood, Florida
  - Wien Center for Memory Disorders, Mount Sinai Medical Center, Miami Beach, Florida
  - Berma Research Group, Plantation, Florida
  - The Roskamp Institute, Sarasota, Florida
  - Comprehensive Neuroscience, Inc., St. Petersburg, Florida
  - Stedman Clinical Trials, LLC, Tampa, Florida
  - USF Memory Disorder's Clinic, Tampa, Florida
  - USF Suncoast Gerontalogy Center, Tampa, Florida
  - Center for Clinical Trials. L.C., Venice, Florida
  - Palm Beach Neurology, West Palm Beach, Florida
  - Lexington Clinic, Lexington, Kentucky
  - Borgess Research Institute, Kalamazoo, Michigan
  - St. Louis University - Clinical Trials Unit, St Louis, Missouri
  - Comprehensive Neuroscience, Inc, Kenilworth, New Jersey
  - Neurological Associates of Albany, PC Neurology, Albany, New York
  - Neurobehavioral Research Inc., Lawrence, New York
  - New York University School of Medicine Aging and Dementia Research Center, New York, New York
  - Columbia University, New York, New York
  - Monroe Community Hospital Program in Neurobehavioral Therapeutics, Rochester, New York
  - Behavioral Medical Research of Staten Island, Staten Island, New York
  - The Ohio State University, Columbus, Ohio
  - Neurology Center of Ohio, Toledo, Ohio
  - Pahl Pharmaceutical Research, LLC, Oklahoma City, Oklahoma
  - Summit Research Network(Oregon) Inc., Portland, Oregon
  - Clinical Trial Specialists, Bala-Cynwyd, Pennsylvania
  - Westmoreland Neurology Associates, Greensburg, Pennsylvania
  - The Clinical Trial Center, LLC, Jenkintown, Pennsylvania
  - Medical University of South Carolina-Alzheimer's Research, Charleston, South Carolina
  - The University of Texas Mental Sciences Instittute, Houston, Texas
  - START Center, San Antonio, Texas
  - Grayline Clinical Drug Trials, Wichita Falls, Texas
  - Southwestern Vermont Medical Center - The Memory Clinc, Bennington, Vermont

RESULTS

PARTICIPANT FLOW:
Groups:
- Donepezil: 5 mg or 10 mg of donepezil hydrochloride (Aricept) taken orally once a day.
Period: Overall Study
Arm/Group | Donepezil | Placebo
Started | 68 | 77
Completed | 55 | 55
Not Completed | 13 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Donepezil | Placebo | Total
Number analyzed (Participants) | 68 | 77 | 145
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.7 (8.46) | 73.4 (8.73) | 72.6 (8.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 36 | 66
  Male | 38 | 41 | 79
Region of Enrollment [Number; unit: participants]
  United States | 68 | 77 | 145

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events
Description: Overview of Treatment-Emergent Adverse Events and Safety Population (TEAEs)
Time Frame: Baseline, Week 6, Week 12 and Week 28.
Measure: Number; unit: Participants
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 68 | 77
Participants
  Any Serious TEAE | 3 | 2
  Any Severe TEAE | 2 | 3
  Any possibly/probably drug-related TEAE | 16 | 32
  Any TEAE causing discontinuation of study drug. | 7 | 17

ADVERSE EVENTS:
Arm/Group | Donepezil | Placebo
Serious Adverse Events (participants affected / at risk) | 3/68 | 2/77
Other Adverse Events (participants affected / at risk) | 11/68 | 20/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Donepezil (N=68) | Placebo (N=77)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pelvic Fracture (Injury, poisoning and procedural complications) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Donepezil (N=68) | Placebo (N=77)
Diarrhea (Gastrointestinal disorders) | 4 | 12
Nausea (Gastrointestinal disorders) | 1 | 7
Abnormal dreams (Psychiatric disorders) | 1 | 5
Insomnia (Psychiatric disorders) | 3 | 5
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 6 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No